CLINICAL TRIAL: NCT00648037
Title: Pilot Trial of Rituximab (Rituxan) for the Prevention of EBV-LPD Post T Cell Depleted Unrelated and HLA Mis-matched Related HSCT
Brief Title: Rituximab (Rituxan) for the Prevention of EBV-LPD Epstein Barr Virus (EBV) Lymphoproliferative Disorder Post T Cell Depleted Unrelated and HLA Mis-matched Related HSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-118
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Hodgkin's Disease; Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma
Keywords: RITUXIMAB; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Leukemia; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Lymphoma | interventions — Rituximab

ARMS (1):
- Rituximab (Experimental): Patients following a T cell depleted HLA-mis-matched related or unrelated hematopoietic stem cell transplant (HSCT) will be treated with monthly Rituximab.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m^2 starting approximately 1 month post transplant (no later than day 45), and continuing monthly until the CD4 cell count is > 200 cells/ul or a maximum of 6 doses have been given.

SUMMARY:
The purpose of this study is to determine if we can prevent Epstein Barr Virus lymphomas by the monthly administration of an (antibody) protein against B lymphocytes called Rituximab. Although this medicine has been approved by the Food and Drug Administration to treat patients with other types of lymphomas, and has been used to treat a small number of patients with EBV lymphomas and other types of B-cell leukemias, it has not been approved to try and prevent EBV-lymphomas. Use of Rituximab to try to prevent EBV-lymphomas is therefore experimental.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be a recipient of aT cell depleted unrelated or HLA mis-matched related HSCT for the treatment of a malignancy or immunodeficiency disease.
* Patients must have an ANC > or = to 1500 cells/ul on the day of first treatment.
* Patients with acute or chronic leukemia, or MDS prior to transplant must be in remission defined as <5% blasts in the bone marrow.
* Patient with must be in remission.
* Patient must be Hepatitis B surface antigen negative pre transplant.
* Patients must have adequate cardiac function defined as a left ventricular ejection fraction at rest of >50% documented pre-transplant.
* Patient may be of either gender and of any ethnic background.
* Patient may be of any age. There is no upper age restriction.
* Patients or their guardians must be able to understand the nature and risk of the proposed study and be able to sign consent.

Exclusion Criteria:

* Karnofsky score <70%
* Female patients who are pregnant or lactating.
* Evidence of EBV-LPD or circulating EBV copy number >1000.
* Active uncontrolled bacterial or fungal infection.
* Prior history of Hepatitis B infection or Hepatitis B surface antigen positivity pre transplant.
* HIV-1,2 sero-positive patients.
* Patients or guardians not signing informed consent.
* Patients with prior allergic reaction to Rituximab or other murine monoclonal antibody.
* Patients taking other investigational agents under another protocol unless discussed and approved in advance by Genentech and the IDEC Therapeutic Director.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trudy Small, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Prophylaxis in TCD Unrelated or HLA Mismatched HSCT: To determine the safety of Rituximab prophylaxis in patients following TCD unrelated or HLA mismatched related HSCT
Period: Overall Study
Arm/Group | Rituximab Prophylaxis in TCD Unrelated or HLA Mismatched HSCT
Started | 26
Completed | 10
Not Completed | 16
Not completed — Not Treated | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 11
Not completed — Relapse | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab Prophylaxis in TCD Unrelated or HLA Mismatched HSCT
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 16
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Safety of Rituximab Prophylaxis
Description: The following stopping rules will be employed to determine that the risks of graft failure, severe GvHD, treatment-related mortality, infection, and EBV-LPD in study patients are not increased over expected. In addition, patients will be removed from study if they develop irreversible non-hematologic Grade III toxicity or any Grade IV toxicity felt to be related or possibly related to study drug.
Time Frame: 3 months post transplant
Population: Please see Adverse Event section for more details.
Measure: Number; unit: participants
Arm/Group | Rituximab Prophylaxis in TCD Unrelated or HLA Mismatched HSCT
Number analyzed (Participants) | 26
participants | 23

ADVERSE EVENTS:
Arm/Group | Rituximab Prophylaxis in TCD Unrelated or HLA Mismatched HSCT
Serious Adverse Events (participants affected / at risk) | 6/26
Other Adverse Events (participants affected / at risk) | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Prophylaxis in TCD Unrelated or HLA Mismatched HSCT (N=26)
Infection w.out neutropenia (Infections and infestations) | 4 (4)
Infection with grade 3/4 neut (Infections and infestations) | 1 (1)
Neutrophils/gran (Infections and infestations) | 1 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Prophylaxis in TCD Unrelated or HLA Mismatched HSCT (N=26)
Alkaline phosphatase (Investigations) | 5 (18)
Bilirubin (Investigations) | 2 (3)
Catheter-rel inf (Infections and infestations) | 4 (4)
Fever (General disorders) | 2 (3)
Hemoglobin (Hgb) (Investigations) | 15 (28)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 7 (9)
Hypotension (Vascular disorders) | 2 (2)
Infection w.out neutropenia (Infections and infestations) | 7 (10)
Leukocytes (Investigations) | 18 (100)
Lymphopenia (Investigations) | 18 (427)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophils/gran (Investigations) | 12 (61)
Platelets (Investigations) | 11 (62)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SGOT (AST) (Investigations) | 5 (7)
SGPT (ALT) (Investigations) | 10 (27)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes